CLINICAL TRIAL: NCT03509740
Title: Efficacy and Safety of Intravenous Tramadol Versus Intravenous Paracetamol for Relief of Acute Pain of Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Intravenous Tramadol Versus Intravenous Paracetamol in Patients With Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Algazeerah hospital (Unknown)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dysmenorrhea
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol (Experimental): Intravenous 100 mg tramadol in 100 ml saline with slow infusion over 10 minutes.
  Interventions: Drug: tramadol
- paracetamol (Active Comparator): Intravenous 1 gm paracetamol in 100 ml saline with slow infusion over 10 minutes.
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: tramadol — 100 mg tramadol in 100 ml saline with slow infusion
  Arms: tramadol
Drug: paracetamol — Intravenous 1 gm paracetamol in 100 ml saline with slow infusion
  Other Names: perfalgan
  Arms: paracetamol

SUMMARY:
Patients presented with primary dysmenorrhea composed the study population. One gram paracetamol and 100 mg tramadol in 100 ml saline with a slow infusion were compared in ceasing dysmenorrhea in the emergency department

DETAILED DESCRIPTION:
Patients over 18 years old who presented with dysmenorrhea composed the study population. Patients received painkiller within the last six hours, physical findings consistent with peritoneal irritation, allergy to the study drugs, renal or liver failure, drug addiction, pregnancy or woman with lactation and denied to give inform consent were the exclusion criteria. The pain of the study patients is measured with the visual analogue scale at baseline, 15th and 30th minutes and 1 hour after study drug administration. At the end of the 60 minutes, rescue drug need is also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe primary dysmenorrhea and visual analog scale (VAS) pain scores ≥40
* Patients over 18 years old

Exclusion Criteria:

* denied to give inform consent, irregular menstrual cycles, known or suspected secondary dysmenorrhea
* Renal or liver failure
* Allergy to the study drugs
* Receiving pain killer within the last 6 hours.
* Physical examination findings consistent with peritoneal irritation
* Pregnancy or patients with lactation
* Drug or Alcohol Abuse

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
acute pain of dysmenorrhea measured by visual analogue scale | 15 minutes
  Change in visual analogue scale at 15th minutes from baseline
pain of dysmenorrhea measured by visual analogue scale | 30 minutes
  Change in visual analogue scale at 30th minutes from baseline
pain of dysmenorrhea measured by visual analogue scale | 60 minutes
  Change in visual analogue scale at 60th minutes from baseline

SECONDARY OUTCOMES:
Rescue drug need | 30 minutes.
  the need for additional analgesic drug
adverse effects. | 60 minutes
  nausea, Vomiting, epigastric pain

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Study Director — Cairo University; mahmoud alalfy, MD, Principal Investigator — National Research Center; Ahmed Ali, mbbch, Principal Investigator — faculty of medicine al-azhar university
Locations (1):
- Aljazeerah Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided